CLINICAL TRIAL: NCT00855907
Title: Prevalence of Fatty Liver in Inflammatory Bowel Disease (IBD) Patients and Mechanisms Related to Inflammation and Fatty Liver
Brief Title: Fatty Liver in Inflammatory Bowel Disease (IBD) Patients
Status: Terminated | Type: Observational
Why Stopped: Lack of budget
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principle investigator - Gastroenterologist, Tel Aviv Sourasky medical center
Other Study IDs: TASMC-09-NM-593-CTIL
Record Dates: First submitted 2009-03-04; First posted 2009-03-05 (Estimated); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Inflammatory Bowel Disease; Fatty Liver
Keywords: IBD; inflammatory bowel disease; fatty liver
MeSH Terms: conditions — Inflammatory Bowel Diseases; Fatty Liver

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood count and biochemistry tests (such as: Liver and thyroid enzimes,cholesterol, immunology, glucose)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cases: IBD patients above the age of 18 years old, suffering from the disease for at least one year.
  Interventions: Other: clinical evaluation

INTERVENTIONS:
Other: clinical evaluation — Patients will fill up a questionnaire regarding their disease, demographic data, other co-morbidities and medications and risk factors for metabolic syndrome.
  Each patient will undergo blood examinations in order to assess inflammation, and metabolic status. Fatty liver will be assessed by liver ultra-sonography.

SUMMARY:
Fatty liver is known to be one of the most frequent liver pathologies in IBD patients (35-40%). Despite this fact, there are only few publications that evaluated the prevalence of fatty liver in IBD patients. Moreover, the pathogenesis of this phenomenon in IBD has not been widely investigated.

The paradox of lean patients and fatty liver can be explained by high use of steroids, by rapid weight loss, and by the abundance of TNFα cytokine in IBD patients that causes insulin resistance.

The aim of the study:

To evaluate the frequency of fatty liver in a cohort of IBD patients and to learn its risk factors.

Methods:

One hundred consecutive IBD patients treated at the Tel Aviv Sourasky Medical Center will be recruited.

Patients will fill up a questionnaire regarding their disease, demographic data, other co-morbidities and medications and risk factors for metabolic syndrome.

Each patient will undergo blood examinations in order to assess inflammation, and metabolic status. Fatty liver will be assessed by liver ultra-sonography.

ELIGIBILITY:
Inclusion Criteria:

* IBD patients above the age of 18 years old, suffering from the disease for at least one year.

Exclusion Criteria:

* Pregnant women,
* Patients suffering from ulcerative colitis after total colectomy,
* HIV patients,
* Patients suffering from other chronic liver disease,
* Patients suffering from cancer currently or in the past, OR
* Patients suffering from any other chronic severe diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: One hundred consecutive IBD patients treated at the Tel Aviv Sourasky Medical Center will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2009-03 (Actual); Primary Completion 2010-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
inflammation and metabolic status | first visit
Assessment of Fatty liver | first visit

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Sourasky Medical center, Tel Aviv, Israel